CLINICAL TRIAL: NCT06267352
Title: Epidemiology and Genomic Surveillance of Methicillin-sensitive Staphylococcus Aureus in ICU Neonatology : Rectal and Nasal Screening, Cross Transmission and Decolonisation
Brief Title: Epidemiology and Genomic Surveillance of Staphylococcus Aureus in ICU Neonatology
Acronym: NEOSAUR
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 230097
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: the Aim of This Study is to Describe Genomic Epidemiology of MSSA in Neonatal ICU
Keywords: cross-transmission; prevention and infection control; bacterial typing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Newborns hospitalized in Neonatology are particularly vulnerable to infections, in particular healthcare associated infection (HAI). Staphylococcus aureus represents the 2nd microorganism responsible for sepsis, this infection is particularly serious and like any HAI, it increases the length of hospitalization of newborns and neonatal morbidity.

In September 2020, the CDC published recommendations for the prevention and control of Staphylococcus aureus infections in neonatal intensive care unit/ICU. They specify the indications for implementing a MSSA surveillance strategy as well as the screening and management methods.

Despite the absence of a defined strategy at the national level, our establishment chose to initiate management measures several years ago following serious infections and MSSA epidemics in neonatal intensive care unit/ICU.

With the aim of improving the efficiency of care and evaluating the strategy chosen at the establishment, it is necessary to describing

* the epidemiology of MSSA carriage and infections
* cross-transmission of MSSA strains between patients
* the success rate of decolonization
* the sensitivity of detection of digestive carriage by stool swabbing in order to limit the number of samples from newborns.

ELIGIBILITY:
Inclusion Criteria:

* newborns hospitalized in neonatal ICU
* MSSA carrier

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MSSA carrier among newborns hospitalized in neonatal ICU
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
frequency of MSSA cross transmission as assessed by WGS | Month 24
  Number of patients with acquired MSSA / total number of MSSA carriers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akinboyo IC, Zangwill KM, Berg WM, Cantey JB, Huizinga B, Milstone AM. SHEA neonatal intensive care unit (NICU) white paper series: Practical approaches to Staphylococcus aureus disease prevention. Infect Control Hosp Epidemiol. 2020 Nov;41(11):1251-1257. doi: 10.1017/ice.2020.51. Epub 2020 Sep 14. No abstract available. PMID 32921340